CLINICAL TRIAL: NCT05802654
Title: Clinical Study of Single Ultra-high Dose Stereotactic Body Radiation Therapy for Early Lung Cancer
Brief Title: Single Ultra-high Dose Stereotactic Body Radiation Therapy for Early Lung Cancer
Acronym: USBRT-1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USBRT-1
Record Dates: First submitted 2023-03-26; First posted 2023-04-06 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Early Lung Cancer; Stereotactic Body Radiotherapy
Keywords: lung cancer; Stereotactic body radiotherapy (SBRT); High dose; Fraction
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: single fraction of ultra-high dose SBRT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants receiving SBRT (Experimental): The participants enrolled will receive single fraction of ultra-high dose SBRT(30Gy/1F).
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — The participants enrolled will receive single fraction of ultra-high dose SBRT(30Gy/1F).

SUMMARY:
The goal of this prospective single-arm phase II study is to study the efficacy and safety of stereotactic body radiotherapy (SBRT) for early lung cancer. The main questions it aims to answer are:

How effective is this regimen of SBRT for early lung cancer? How safe is this regimen of SBRT for early lung cancer?

DETAILED DESCRIPTION:
The goal of this prospective single-arm phase II study is to study the efficacy and safety of stereotactic body radiotherapy (SBRT) for early lung cancer. This study intends to enroll 100 participants in 2 years. The participants enrolled will receive single fraction of ultra-high dose stereotactic body radiotherapy (SBRT) (30Gy/1F).

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent;
2. Male or female aged ≥ 18 years and ≤ 75 years;
3. patients with early stage lung cancer confirmed by pathology or clinical MDT;
4. The physical state score (ECOG PS) of the eastern tumor cooperative group was 0 ~ 1;
5. Expected survival time ≥3 months;
6. Laboratory results during screening must meet the following requirements:

   1. Blood routine: neutrophil absolute count (ANC) ≥ 1.5 × 109/L, platelet count (PLT) ≥ 100 × 109/L, hemoglobin (HGB) ≥ 90 g/L (no blood transfusion or erythropoietin dependence within 7 days);
   2. Liver function: total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal value (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) were less than 2.5 times ULN in subjects without liver metastasis, and ALT and AST were less than 5 times ULN in subjects with liver metastasis.
   3. Renal function: serum creatinine (Cr) ≤1.5 times ULN or Cr clearance ≥60 mL/min (Cockcroft-Gault formula), and urine protein (UPRO) &lt on routine urine test; 2+ or 24 h urinary protein quantification < 1g;
   4. International standardized ratio (INR) ≤1.5 times ULN and partial prothrombin time (PTT) or activated partial thrombin time (APTT) ≤1.5 times ULN during the 7 days prior to treatment;
7. For female subjects of reproductive age, urine or serum pregnancy tests should be negative within 3 days prior to receiving the first fraction of SBRT. If the urine pregnancy test results cannot be confirmed negative, a blood pregnancy test is requested;
8. Compliance with the research protocol is expected to be good.

Exclusion Criteria:

1. currently participating in an interventional clinical trial;
2. any unstable systemic disease, including but not limited to active infection, congestive heart failure [New York Heart Association (NYHA) class ≥ II], severe arrhythmia requiring medical therapy, liver, kidney, or metabolic disease; Type I and type II respiratory failure;
3. other malignancies within 5 years before randomization, except adequately treated cervical carcinoma in situ, basal cell or squamous skin cancer, local prostate cancer after radical surgery, ductal carcinoma in situ after radical surgery, or papillary thyroid cancer;
4. women who are pregnant or breastfeeding or who plan to become pregnant or breastfeeding during the study period;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
PFS | 3 years
  The time from the date of treatment to the date of disease progression or death or last follow-up.

SECONDARY OUTCOMES:
OS | 3 years
  The time from the date of treatment to the date of death or last follow-up.
AE | 3 years
  The incidence of All adverse event (AE), treatment emergent AE (TEAE), treatment-related AE (TRAE), immune-related AE (irAE), serious AE (SAE) and radiation-related AE(rAE), the relevance and severity related with the study protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Hongqing Zhuang, M.D., Study Chair — Department of Peking University Third Hospital
Locations (1):
- Department of radiation oncology, Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Statistical Analysis Plan, and Clinical Study Report will be shared with researchers for research use after permission was obtained from the study institution.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 6 months after publication
Access Criteria: Researchers